CLINICAL TRIAL: NCT01713660
Title: A MULTI-CENTER PROSPECTIVE STUDY TO EVALUATE THE USE OF THE INTRALASE iFS™ FEMTOSECOND LASER SYSTEM TO CREATE CLEAR CORNEAL INCISIONS AND PARACENTESIS INCISIONS FOR CATARACT SURGERY
Brief Title: Corneal Incisions With the IntraLase iFS Femtosecond Laser System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMTO-105-CCIP
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Results first posted 2013-05-29 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cataract
Keywords: Cataract surgery; Femtosecond laser; Corneal incisions
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FS Corneal Incisions (Other)
  Interventions: Device: iFS Femtosecond Laser

INTERVENTIONS:
Device: iFS Femtosecond Laser — corneal incisions created by the femtosecond laser

SUMMARY:
The IntraLase iFS femtosecond laser system can create corneal arcuate incisions for cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Unilateral or bilateral cataract(s) for which phacoemulsification lens extraction and posterior chamber intraocular lens (IOL) implantation has been planned
* Visual potential of 20/25 or better in each study eye following cataract removal and IOL implantation
* Clear intraocular media other than cataract
* Available, willing and capable of complying with examination procedures and follow-up visits for the duration of the study
* Signed informed consent

Exclusion Criteria:

* Previous intraocular or corneal surgery, including refractive surgery in the operative eye(s)
* History of active or recurrent ophthalmic disease
* Abnormal topography, including evidence of keratoconus or pellucid marginal degeneration or irregular astigmatism in the operative eye(s)
* White to white measurement less than 10 mm or greater than 14 mm
* Corneal pathology/abnormality that may interfere with the transmission of laser energy, laser light or precludes applanation
* Corneal pathology/abnormality that is predicted to cause visual acuity losses to a level of 20/30 (Snellen) or worse during the study
* Subjects with diagnosed degenerative visual disorders (e.g., macular or other retinal pathology) that are predicted to cause visual acuity losses to a level of 20/30 (Snellen) or worse during the study
* Subjects with conditions associated with increased risk of IOL/capsule instability
* Pharmacologically dilated pupil size less than 5.5 mm or the presence of any pupil abnormalities
* Prior, current, or anticipated use during the course of the study of tamsulosin, silodosin or pilocarpine (e.g. Flomax, Flomaxtra, Rapaflo)
* History of any ocular or medical conditions that could affect corneal wound healing
* Poorly-controlled diabetes or subjects with diabetic retinopathy
* Concurrent use of topical or systemic medications that may impair corneal wound healing
* Acute, chronic, or uncontrolled systemic or ocular disease or illness that would, in the opinion of the investigator, increase the operative risk or confound the outcome(s) of the study (e.g., immunocompromised, connective tissue disease, etc.)
* Ocular hypertension (> 21 mm Hg)
* Women who are pregnant, breast-feeding, or intend to become pregnant over the course of the study
* Known sensitivity or inappropriate responsiveness to any of the medications used in the post operative course
* Concurrent participation or participation in any other clinical trial during the duration of this clinical study including 30 days prior to preoperative visit

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from private medical practices from October to December 2012
Pre-assignment Details: No preassignment details
Groups:
- FS Corneal Incisions: iFS Femtosecond Laser : corneal incisions created by the femtosecond laser
Period: Overall Study
Arm/Group | FS Corneal Incisions
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FS Corneal Incisions
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Demonstration That the Femtosecond Laser Consistently Produces Desired Incisions.
Description: Evaluation of incisions created as programmed and measurement in mm. Data reported will be based on intended incision size (as programmed) vs. achieved incision size (as measured).
Time Frame: Day 0, Operative (Within 2 hours of incision creation)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | FS Corneal Incisions
Number analyzed (Participants) | 37
Number analyzed (eyes) | 37
mm
  Achieved Clear Corneal Incision (CCI) Measurement | 2.75 (0.09)
  Intended CCI Incision Size (as programmed) | 2.74 (0.08)

2. Secondary Outcome: Surgeon Assessment of Workflow
Description: Surgeon questionnaire (completed at the end of each surgery and the end of each surgical day): Were incisions created as intended?
Time Frame: Day 0, Operative
Measure: Number; unit: percentage of yes answers
Arm/Group | FS Corneal Incisions
Number analyzed (Participants) | 37
percentage of yes answers | 97.3

3. Secondary Outcome: Percent of Seidel Staining
Description: Demonstration of no wound leakage as measured by Seidel test at slit lamp with fluorscein dye. A negative Seidel test result indicates no wound leakage.
Time Frame: Day 0 (performed immediately post-incision creation), Day 1
Measure: Number; unit: percentage of eyes with negative Seidel
Units Other Than Participants: eyes
Arm/Group | FS Corneal Incisions
Number analyzed (Participants) | 37
Number analyzed (eyes) | 37
percentage of eyes with negative Seidel | 100

ADVERSE EVENTS:
Time Frame: The time frame for reporting adverse event reports was 1 month.
Arm/Group | FS Corneal Incisions
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement including "Neither Institution nor Principal Investigator shall have any right to publish or present any information or results concerning the Study without express written consent of Sponsor. Under no circumstances shall Institution or Principal Investigator publish or disclose any of Sponsor's proprietary information, as defined by the CDAs, without Sponsor's prior written approval."